CLINICAL TRIAL: NCT04595071
Title: Functional Outcomes of Voice Recognition Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberating Technologies, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 120180305; 1R43HD095750-01 (NIH); 120180305 (Other: NEIRB)
Record Dates: First submitted 2020-09-25; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Prosthesis; Amputation; Prosthesis User
Keywords: voice recognition; prosthetics; upper limb

STUDY DESIGN:
Intervention Model Description: Voice-Activated Prosthesis Interface
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Control (No Intervention): Use of standard two-site myoelectric control of multi-articulating hand.
- Voice Recognition Control (Experimental): Use of voice recognition control in addition to standard two-site myoelectric control of a multi-articulating hand.
  Interventions: Device: Voice Activated Prosthetic Interface (VAPI) Controller

INTERVENTIONS:
Device: Voice Activated Prosthetic Interface (VAPI) Controller — A device installed between a subjects socket quick disconnect wrist connection and multi-articulating hand which enables the use of voice as a control modality in addition to their standard two-site myoelectric control.
  Arms: Voice Recognition Control

SUMMARY:
The purpose of this study is to evaluate the use of a voice activated prosthesis interface controller for functional outcomes as compared to standard prosthesis control.

DETAILED DESCRIPTION:
The study will take place over two separate visits spaced about 1 week apart.

During the first visit participants will undergo informed consent. They will then be randomly assigned one of two test conditions, (a) standard control, or (b) voice recognition control.

For both conditions participants will be allowed to train on the control scheme until they are comfortable with it's usage. Subjects will then be asked to manipulate common objects as a test of improved control and utility. Functional outcome measures will be utilized to standardize the tasks performed and evaluate the advantages of voice control.

On the second visit participants will be assigned the alternate condition, allowed to train with the control scheme, and run through the same set of functional outcomes measures.

Upon completion of the second visit participants will be asked to fill out a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Be willing and able to complete the tasks outlined in the study
* Are at least 6 months post amputation
* Have used an upper limb myo-prosthesis
* Necessary prosthesis components to interface to the proposed device
* Have no injury to the residual limb or shoulder that will impact their participation in this study
* Must be current users of upper limb myo-prosthesis or able to wear a prosthesis simulator brace
* Users who utilize multi-articulating hand terminal devices, and specifically Touch Bionics iLimb or Steeper beBionic hand users will be preferred, as these are the targeted devices that will be used during testing.
* Subjects must also be able to speak English in order to be properly consented as well as to interface with the voice recognition module (only English will be included in this feasibility study).

Exclusion Criteria:

* The risks to pregnant people and fetuses are unknown and therefore pregnant people should not participate in the study and will be screened by self-disclosure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
University of New Brunswick (UNB) Test of Prosthetics Function | 2 Days
  A Test for Unilateral Upper Limb Amputees

SECONDARY OUTCOMES:
Custom Activities of Daily Living (ADL) Tasks | 2 Days
  Timed completion of a set of custom ADL
Grip Switch Assessment (GSA) | 2 Days
  Timed completion of a randomized set of multi-articulating hand grip switches

OTHER OUTCOMES:
Missed grips | 2 Days
  A count of the number of intended missed grip changes

CONTACTS AND LOCATIONS:
Locations (1):
- Liberating Technologies, Inc., Holliston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNB Test of Prosthetics Function — https://www.unb.ca/research/institutes/biomedical/_resources/docs/unb_test_of_prosthetics_function.pdf

DOCUMENTS (1):
  • Informed Consent Form (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT04595071/ICF_000.pdf